CLINICAL TRIAL: NCT01042366
Title: Randomized Phase II Evaluation of Immunization Against Tumor Cells in Subjects With Metastatic Melanoma Using Autologous Mature Dendritic Cells
Brief Title: Dendritic Cells (DC) Vaccine for Metastatic Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed to accrual in March 2009 for slow accrual.
Sponsor: John Kirkwood (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Kirkwood, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 01-171; 5P01CA073743 (NIH)
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine co-cultured with melanoma cells (Experimental): Dendritic Cells co-cultured with melanoma cells injected as a vaccine intra/peri-nodally under ultrasound guidance
  Interventions: Biological: Vaccination
- Vaccine pulsed with tumor cell lysates (Experimental): Dendritic Cells pulsed with tumor cell lysates were injected as a vaccine intra/peri-nodally under ultrasound guidance
  Interventions: Biological: Vaccination
- Vaccine fused with tumor cells (Experimental): Dendritic Cells fused with tumor cells were injected as a vaccine intra/peri-nodally under ultrasound guidance
  Interventions: Biological: Vaccination

INTERVENTIONS:
Biological: Vaccination — Subjects will receive as an outpatient 4 weekly ultrasound-guided intra/peri-lymph nodal administrations of the autologous tumor dendritic cell vaccine. The dose of the autologous tumor cell dendritic cells/vaccine will be 1-5 X 106.

SUMMARY:
The purpose of this study is to determine what effect using an experimental tumor vaccine (a substance or group of substances meant to cause the immune system to respond to a tumor) made using patients' own tumor cells and blood cells will have on their melanoma.

DETAILED DESCRIPTION:
Historically, metastatic melanoma has been associated with a poor prognosis. Recently, numerous immunotherapeutic agents, particularly checkpoint inhibitors, have moved to the forefront of therapy. Checkpoint inhibitors such as ipilimumab, pembrolizumab, and nivolumab have revolutionized the treatment of melanoma. Despite this, not all patients respond to checkpoint inhibitors, and even patients who initially respond to checkpoint inhibitor therapy often later relapse (median response duration of 2 years); complete responses remain uncommon. Thus, more effective immunotherapies are clearly needed.

The concept of administering dendritic cell (DC)-based vaccines to prompt an immune response against tumor cells has shown promise in the treatment of advanced cancers. Sipuleucel-T, now FDA-approved for the treatment of advanced prostate cancer, is one such vaccine that consists of autologous antigen-presenting cell (APC) activated ex vivo by a fusion protein consisting of the antigen prostatic acid phosphatase (PAP) and granulocyte-macrophage colony stimulating factor (GM-CSF). Although response rates to Sipuleucel-T are low, recent studies suggest that DC vaccines have the potential to improve survival by increasing the breadth and diversity of melanoma-specific T cells.

It is known that the method of antigen (Ag) delivery is important for the success of DC vaccines, but it remains unclear which method is most effective in producing antitumor responses. Approaches tested clinically include pulsing with HLA-restricted defined peptide Ags, loading with purified proteins, transfecting with mRNA, engineering with Ag-encoding viral vectors, and using autologous tumor cells or allogeneic cell lines directly as sources of Ag. Efficacy can be measured in vivo using surrogate endpoints, such as development of tumor-specific delayed-type hypersensitivity (DTH) reactions. Prolonged survival of vaccinated melanoma patients has been reported to correlate with induction of positive DTH tests. Antitumor activity may also be assessed by ELISpot analysis of the frequency of tumor-Ag specific IFNγ-producing T cells. To assess the quality of the DC vaccines, surrogate markers of DC function including maturation markers, co-stimulatory molecule expression, and IL12p70 production, a critical cytokine in antitumor response, can be measured

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have Stage III-IV melanoma (any tumor thickness and any number of lymph node involvement, and in-transit metastases, or distant metastases) (AJCC). Each diagnosis will be confirmed by pathology review at the Melanoma Center of the University of Pittsburgh Cancer Institute.
* All subjects have to be HLA-A2 positive (required for immunologic testing).
* Subjects must have recovered fully from surgery.
* Availability of resectable or tissue banked tumor cells for autologous tumor dendritic cell vaccine preparation.
* Sufficient number of tumor cells available for autologous tumor dendritic cell vaccine preparation (min 2.6 x 10 7).
* Sufficient number of DCs of at least 12 X 10 6 for preparation of the autologous tumor dendritic cell vaccine preparation (if less than needed number of cells will be obtained by one course of leukopheresis, the second leukopheresis will be repeated 2 weeks apart).
* Subjects must not have received any chemotherapy or immunotherapy within the four weeks preceding vaccination (six weeks for nitrosourea, mitomycin).
* Subjects must have an expected survival of greater than or equal to 12 months.
* Subjects must have an ECOG performance status 0 or 1.
* Subjects must have the following initial and subsequent pretreatment
* laboratory parameters: Granulocytes >=2,500/mm3 Lymphocytes >=1000/mm3 Platelets >100,000/mm3 Serum Creatinine <=1.5 X the ULN AST, ALT, GGT, LDH, Alk phos <= 2.5 X the ULN Serum Bilirubin <=1.5 X ULN
* Subjects must be >= 18 years of age and must be able to understand the written informed consent.
* No evidence of active infection, regardless of the degree of severity or localization. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.
* Subjects with measurable disease must have an evaluation for extent of disease (tumor staging) performed within 30 days of start of treatment.
* Pretreatment baseline evaluations for laboratory parameters must be obtained within 10 to18 days of subject registration

Exclusion Criteria:

* Subjects currently treated with anti inflammatory agents including glucocorticoid therapy are ineligible.
* Subjects currently on treatment with steroids are ineligible, but may receive the DC autologous tumor dendritic cell vaccine 4 weeks after steroid cessation. Subjects on maintenance steroids because of adrenal insufficiency are eligible.
* Subjects with severely abnormal liver function tests [AST (SGOT), ALT (SGPT), GGT, Alk.Phos, LDH, and total bilirubin greater than 2 X ULN].
* Subjects with uncontrolled pain.
* Subjects with autoimmune disease, HIV, and hepatitis
* Subjects with symptomatic brain metastasis.
* Subjects with active prior malignancy (with exception of non-melanoma skin cancers and carcinoma in situ of the cervix).
* Subjects who have been previously immunized with melanoma vaccine until 10 subjects have been registered in each treatment arm.
* Subjects who are pregnant.
* Subjects who have sensitivity to drugs to provide local anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Kirkwood, MD, Principal Investigator — UPMC UPCI HCC
Locations (1):
- Upmc Upci Hcc, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 16 subjects were enrolled, one subject was referred to hospice and never began the study.
Groups:
- DCs Co-cultured With Melanoma Cells: DCs co-cultured with melanoma cells
  Vaccination: Subjects will receive as an outpatient 4 weekly ultrasound-guided intra/peri-lymph nodal administrations of the autologous tumor dendritic cell vaccine. The dose of the autologous tumor cell dendritic cells/vaccine will be 1-5 X 106.
  Leukapheresis: All selected subjects will undergo leukapheresis. Two and a half times the subject's blood volume will be processed per procedure. A single 4 hour leukapheresis will be done.
- DCs Pulsed With Tumor Cell Lysates: DCs pulsed with tumor cell lysates
  Vaccination: Subjects will receive as an outpatient 4 weekly ultrasound-guided intra/peri-lymph nodal administrations of the autologous tumor dendritic cell vaccine. The dose of the autologous tumor cell dendritic cells/vaccine will be 1-5 X 106.
  Leukapheresis: All selected subjects will undergo leukapheresis. Two and a half times the subject's blood volume will be processed per procedure. A single 4 hour leukapheresis will be done.
- DCs Fused With Tumor Cells: DCs fused with tumor cells
  Vaccination: Subjects will receive as an outpatient 4 weekly ultrasound-guided intra/peri-lymph nodal administrations of the autologous tumor dendritic cell vaccine. The dose of the autologous tumor cell dendritic cells/vaccine will be 1-5 X 106.
  Leukapheresis: All selected subjects will undergo leukapheresis. Two and a half times the subject's blood volume will be processed per procedure. A single 4 hour leukapheresis will be done.
Period: Overall Study
Arm/Group | DCs Co-cultured With Melanoma Cells | DCs Pulsed With Tumor Cell Lysates | DCs Fused With Tumor Cells
Started | 5 | 6 | 4
Completed | 5 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DCs Co-cultured With Melanoma Cells | DCs Pulsed With Tumor Cell Lysates | DCs Fused With Tumor Cells | Total
Number analyzed (Participants) | 5 | 6 | 4 | 15
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 72] | 44.5 [32 to 59] | 54 [49 to 81] | 49 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Delayed Type Hypersensitivity (DTH) Response
Description: Delayed type hypersensitivity (DTH) response to antigen-loaded autologous, dendritic cell vaccine (DC) injected intradermal in vivo
Time Frame: 12 mo
Population: Patients who met inclusion criteria and received at least 3 doses of the vaccine
Measure: Number; unit: participants
Arm/Group | DCs Co-cultured With Melanoma Cells | DCs Pulsed With Tumor Cell Lysates | DCs Fused With Tumor Cells
Number analyzed (Participants) | 5 | 6 | 4
participants | 2 | 2 | 1

2. Primary Outcome: ELISpot Response to Melanoma
Description: Peripheral blood CD8+ and CD4+ T cell responses against autologous tumor cells, and HLA-presented melanoma epitopes, using ELISPOT and MHC-peptide tetramer assays.
Time Frame: 12 mo
Population: Patients who met inclusion criteria and received at least 3 doses of the vaccine
Measure: Number; unit: participants
Arm/Group | DCs Co-cultured With Melanoma Cells | DCs Pulsed With Tumor Cell Lysates | DCs Fused With Tumor Cells
Number analyzed (Participants) | 5 | 6 | 4
participants | 2 | 2 | 1

ADVERSE EVENTS:
Description: Adverse events were not collected/monitored per Arm/Group
Groups:
- All Participants (Overall Study): For all arms: DC vaccine Co-cultured With Melanoma Cells; DC Vaccine Pulsed With Tumor Cell Lysates; DC Vaccines Fused With Tumor Cells
Arm/Group | All Participants (Overall Study)
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=15)
Hepatic-Other (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (Overall Study) (N=15)
Hemoglobin (Blood and lymphatic system disorders) | 4
Platelets (Investigations) | 1
Edema (General disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 4
Constitutional Symptoms-Other (General disorders) | 3
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 1
Flushing (Vascular disorders) | 1
Injection site reaction (General disorders) | 5
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Diarrhea patients without colostomy (Gastrointestinal disorders) | 1
Dyspepsia/heartburn (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 1
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 1
Hepatic-Other (Hepatobiliary disorders) | 2
Alkaline phosphatase (Investigations) | 1
Infection (documented clinically or microbiologically) with grade 3 or 4 neutropenia (Infections and infestations) | 1
Lymphatics-Other (Blood and lymphatic system disorders) | 1
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Neurology-Other (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Dizziness/lightheadedness (Nervous system disorders) | 1
Mood alteration-anxiety, agitation (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathic pain (Nervous system disorders) | 1
Mood alteration-depression (Psychiatric disorders) | 1
Neuropathy-sensory (Nervous system disorders) | 3
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pain-Other (General disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes